CLINICAL TRIAL: NCT05618730
Title: Safety, Tolerability, Plug Retention and Preliminary Efficacy of Tacrolimus-loaded Punctal Plug in Patients With Moderate to Severe Dry Eye Disease - Cohort B
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eximore Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXP-TC-1
Record Dates: First submitted 2022-11-03; First posted 2022-11-16 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Dry Eye; Keratoconjunctivitis Sicca; Ocular Inflammation
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca | interventions — Lubricant Eye Drops

STUDY DESIGN:
Intervention Model Description: Each patient with Dry Eye Disease is tested with EXP-TC tacrolimus releasing punctal plug in one eye. Both eyes will receive standard of care of 0.15% sodium hyaluronate (Hyabak, Théa laboratories).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXP-TC punctal plug together with artificial tears (Experimental): EXP-TC: A punctal plug as a delivery system for Tacrolimus. EXP-TC has 3 different sizes (Small, Medium and Big for Wide EXP-TC)
  Interventions: Device: punctum plug insertion; Drug: Eye Drops, Lubricant
- Artificial tears (Active Comparator): Preservative-free, 0.15% sodium hyaluronate (Hyabak, Théa laboratories)
  Interventions: Drug: Eye Drops, Lubricant

INTERVENTIONS:
Device: punctum plug insertion — EXP-TC delivers the anti-inflammatory drug tacrolimus that acts as inhibitor of T lymphocytes and may therefore lead to the inhibition of release of inflammatory cytokines.
  EXP-TC has a Pangolin design and has 3 different designs: big, medium and small with drug content ranging from 194 to 348 µg.
  After plug insertion preservative-free, 0.15% sodium hyaluronate (Hyabak, Théa laboratories) is taken 4 times daily.
  Arms: EXP-TC punctal plug together with artificial tears
Drug: Eye Drops, Lubricant — Preservative-free, 0.15% sodium hyaluronate (Hyabak, Théa laboratories) 4 times daily.

SUMMARY:
The purpose of this interventional study is to assess safety, patient tolerability, plug retention rate, and preliminary efficacy in improving the symptoms of Dry Eye Disease (DED) of EXP-TC tacrolimus releasing punctal plug. The main questions it aims to answer are:

1. The safety of using EXP-TC plug following all study adverse events
2. The number of patients with Adverse Events related to the us of EXP-LP plug
3. The number of patients discontinuing the study due to plug discomfort
4. The total patients with plugs remained during the 3-months study duration from plug insertion
5. Exploratory: change from baseline in the study eye to follow-up visits in various Dryness clinical measurements. The change of measurements from baseline will also be compared between the study and fellow control eye (receiving artificial tears only, 0.15% sodium hyaluronate).

DETAILED DESCRIPTION:
Device Description - EXP-TC punctual plug is a delivery system for Tacrolimus- an immunosuppressive macrolide drug that is has been proved to improve Dry-Eye Disease (DED) symptoms, similar to and sometimes better than the well-known cyclosporine. The EXP-TC punctual plug is designed for insertion into the punctual opening. The plug is molded of a medical-grade composite containing Tacrolimus. The plug design features a flattened head/rim which remains outside the punctum and a central neck/shaft which tapers outward toward a nose. The plug is designed to create a vector force to keep the plug snugly in the punctual opening. As soon as the tears wet the plug, the drug is locally released. The plug has Pangolin design with 3 different sizes, Small, Medium and Big.

The commercial lubricant (positive study control) preservative-free, 0.15% sodium hyaluronate (Hyabak) is marketed by, Théa laboratories and is known as a common first-line treatment for DED

Study Design - This is a prospective, single center, open-label, self-controlled ("split body" design) non-randomized single eye study performed on patients with moderate to severe dry eye disease.

Study Population and Justification - Up to 20 patients with DED in both eyes will be enrolled. Due to early feasibility stage of the study, no formal sample size calculation was done for this study.

The intent to treat (ITT) population, defined as enrolled participants not including those who leave the study prematurely during the screening period (before EXP-TC insertion).

Handling of Participant Withdrawals - participants who leave the study prematurely during study will not be replaced. The discontinuing patient will be followed for safety by a phone call, one month after exiting the study. Each case of premature withdrawal will be properly recorded.

Patient Screening - Prior to any study-related procedure, delegated study team members will approach potentially eligible adult subjects diagnosed with moderate to severe dry eye disease. Those who may be eligible will be offered the choice of undergoing screening to be enrolled in the study or receiving standard public treatment for their current illness without participating in the study. Subjects who do not meet inclusion criteria or who are for any other reason determined to be too ill for inclusion in the study, or who decline to participate in the study, will be considered and recorded as "screen failure" and receive standard and appropriate treatment.

Informed Consent: The informed consent document will be signed and dated for screening and enrollment and each patient consenting will be documented in the patient medical binder. The patient will be given a copy of the consent form together with the study doctor's letter at the time of enrollment. The clinician will ask the patient about his plans and his willingness to attend all scheduled follow-up visits.

Each patient is considered as a Block unit with one studied eye and contra lateral fellow eye. Patients will be identified by a serial number and will be numbered according to their serial recruitment (3 digits).

TRIAL PROCEDURES:

Patients will be identified and offered to be enrolled in the study during a routine clinic visit.

After informed consent is obtained, an electronic case record form (eCRF) including all aspects listed below will be recorded. Eligible patients will be enrolled into the study and will be monitored according to ophthalmic standard examinations (see below).

Visit 1: Screening and washout (2 weeks before EXP-TC plug insertion) During the screening visit, patients will be offered to participate in the study and sign an informed consent. An immunologist lab test diagnosing Sjogren's syndrome would be requested from all screened patients.

Afterward, inclusion and exclusion criteria will be verified. Assessments will include Dryness visual analog scale (VAS), a complete eye exam which will comprise: Best-corrected visual acuity (BCVA), biomicroscopic examination including dilated fundus examination, non-invasive (NIKBUT) and fluorescein tear break-up time (TBUT), and Corneal staining with fluorescein and grading according to NEI corneal fluorescein staining (CFS) score. Central Corneal Thickness (CCT), and Schirmer test type I will also be evaluated. The Schirmer strip will be frozen at -20oC for future PK determination.

There will be pre-enrollment washout of all eye-drop medications for a duration of 2 weeks from study inclusion. During that time 0.15% sodium hyaluronate (Hyabak, Théa laboratories) will be administrated to both eyes 4 times daily. Therefore, subjects will be discharged after being instructed to stop using all relevant medications for 2 weeks.

Visit 2: Day 0, Investigational EXP-TC plug insertion:

Eligibility will be reconfirmed. Assessments will include: Dryness visual analog scale (VAS), Ocular Discomfort Score (ODS), TBUT and NIKBUT. A complete eye exam will include: Best-corrected visual acuity (BCVA), Anterior Segment Exam, biomicroscopic examination, Corneal staining with fluorescein and grading according to NEI corneal fluorescein staining (CFS) score. Lissamine green staining, Central Corneal Thickness (CCT), Schirmer test type I, and IOP will also be evaluated. The Schirmer strip will be frozen at -20oC for future PK determination.

One eye will be chosen as the study eligible eye. If both eyes are considered eligible, the eye with the higher staining CFS scores or with the lower Schirmer result (more severe) will be selected as the study eye. If insertion is unsuccessful, the fellow eligible eye (even if less severe but still eligible) can be considered the study eye with the EXP-TC plug inserted.

Before punctual plug placement, the lacrimal duct anatomy will be assessed using Katena Products Inc. - Coroneo punctual gauge Using the physician biomicroscope, a suitable-size EXP-TC punctual plug will be initially inserted in the lower punctum on the side of the study eye using standard curved forceps under topical anesthesia following topical prophylactic antibiotics. It is recommended to lubricate the plug with sterile saline solution or artificial tears to ease insertion. Another plug size will be inserted if unsuccessful (due to technical difficulty or inconvenience to the patient). The location and stability of the implant will be verified and documented.

Patients will be discharged home and asked NOT to take any eye drops in both eyes except the standard of care of 0.15% sodium hyaluronate (Hyabak, Théa laboratories) 4 times daily throughout the follow-up.

Visits 3, 4, 5, 6, 7: Follow-up visits Following visits will be on days 2, 7, and on weeks 2, 4, and 6 after plug insertion.

Assessments will include Dryness visual analog scale (VAS), Ocular Discomfort Score (ODS), Oculus keratography for Tear breakup time (NIKBUT) and tear break-up time (TBUT). A complete eye exam will include Best-corrected visual acuity (BCVA), Anterior Segment Exam, biomicroscopic examination, Corneal staining with fluorescein, and grading according to NEI Corneal Fluorescein Staining (CFS) score. Lissamine green staining, Central Corneal Thickness (CCT) and Schirmer test type I will also be evaluated. The Schirmer strip will be frozen at -20oC for future PK determination.

*Visit 4 (7 days after plug insertion): In compliance with the Centric Patient Approach, delegated study member will call the patient facility on the specific day scheduled together. The patient will be asked to report any insertion or post-insertion complication (e.g.) - all will be investigated by the study nurse using the safety Follow Up Form. In addition, the patient will be asked for any other non-ophthalmic Adverse Events and any change in Concomitant medications. A detailed description of the study procedures to be performed in each visit is included in Table 1 below - Procedure per Visit.

The placement of the plug will be verified. If the plug is not visualized or the patient complains of discomfort that the investigator believes is related to the plug, the investigator can choose to insert another plug up to a maximum of 3 successful replacements (a maximum of four plugs). A plug replacement will be considered only after it was successfully inserted in the punctum following visit discharge. The EXP-TC plug that has been removed should be stored at -20 Celsius for future analysis.

Termination visit - the investigator will remove the EXP-TC medicated punctual plug using routine curved eye forceps. The EXP-TC plug will be stored at -20 Celsius for future analysis. Dilated fundus exam would also be done. The patient will be discharged home with eye medication as needed, prescribed by the study investigator for both eyes.

Un-scheduled visit/s:

The study investigator will instruct the patient to immediately contact the study team in case of any of those: plug loss, intraocular inflammation, eyelid edema and keratitis.

The patient must call the study nurse to schedule an un-scheduled visit which may only be performed by one of the study investigators, and will be reported to the principal investigator. In such cases, an un-scheduled visit form will be filled out. For unscheduled visits the patient will be clinically managed by the study team with additional eyes examination to be done at the discretion of the investigator.

Data Monitoring and Quality Control - The investigator, through an appointed Clinical Research Associate (CRA), will be responsible for implementing and maintaining quality assurance and quality control systems with written Standard Of Procedures to ensure that trials are conducted and data are generated, documented (recorded), and reported in compliance with the protocol, GCP, and the applicable regulatory requirement(s), including ISO 14155:2020.The investigator will be responsible for ensuring direct access to all trial related sites, source data/documents, and reports for the purpose of monitoring and auditing by the hospital, and inspection by Israeli regulatory authorities. Quality control should be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly. The study CRA will verify that (a) The rights and well-being of human patients are protected, (b) The reported trial data are accurate, complete, and verifiable from source documents and (c) The conduct of the trial is in compliance with the currently approved protocol/amendment(s), with GCP, and with the applicable regulatory requirement(s) (including ISO 14155:2020). The monitor will submit a written report after each trial-site visit or trial related communication. A report should include the date, site, name of the monitor, and name of the investigator or other individual(s) contacted. A report should include a summary of what the monitor reviewed and the monitor's statements concerning the significant findings/facts, deviations and deficiencies, conclusions, actions taken or to be taken and/or actions recommended to secure compliance. To ensure compliance of this investigator initiated trial with current national regulations and the ICH guidelines, data generated by this study will be available for inspection upon request by representatives of the local health authorities- IRB or the national authorities - MOH, or any entity providing support for this trial. The general scope of such visits would be to inspect study data (regulatory requirements), source documentation and CRF completion in accordance with current GCP, the ICH guidelines and the respective local and national government regulations and guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age and over;
2. Patient-reported history of DED in both eyes
3. Use of artificial tears within 3 months before the Screening Visit
4. Corneal fluorescein staining score ≥2 (0- to 4-point scale) in ≥1 region (superior, inferior, or central) in at least one eye
5. Schirmer ≥1 and ≤10 mm in both eyes
6. Central corneal thickness of 400-620 microns.
7. IOP ≤ 24 mmHg in each eye

Exclusion Criteria:

1. Intolerance or contraindication to Tacrolimus
2. Stevens-Johnson Syndrome;
3. Use of methotrexate or systemic cyclosporine within the 3 months before the Screening Visit;
4. Using systemic anti-rheumatic therapy, if started within 6 months before recruitment OR that the systemic disease is considered unstable OR that the patient is unsure of continuing using the treatment throughout the current study;
5. Use of any anti-rheumatic biological agent within 2 months, or 5 half-lives, whichever is longer, before the Screening Visit;
6. Use of oral corticosteroids >10 mg prednisone, or equivalent, per day, if started within 2 months before screening;
7. Use of topical steroids within 4 weeks before the Screening Visit and for the duration of the study
8. Use of oral statin or preparation containing omega-3 fatty acid unless dose has been stable for at least 3 months and will remain so during the trial;
9. Presence of chronic ocular disease other than Aqueous-Deficient Dry Eye requiring topical treatment.
10. Presence of post-burn ocular injury;
11. Active ocular herpes simplex virus infection;
12. Concomitant use of contact lenses or use within 3 months before the Screening Visit or inability to abstain from contact lens use throughout the study.
13. Persistent intraocular inflammation or infection;
14. Have anterior blepharitis, which is deemed clinically significant and likely to interfere with study parameters in the opinion of the investigator;
15. Meibomian gland dysfunction (MGD) necessitating treatment in the 4 weeks before or planned during the study period.
16. Surgical occlusion of the lacrimal puncta, including the insertion of punctual plugs, within 3 months of the Screening
17. Continuous cough OR fever/high temperature (38.0oC or greater) OR loss of/change in the sense of smell or taste (anosmia).
18. Recent ocular or eyelid surgery
19. Pregnant women or women suspected of being pregnant, nursing mothers
20. Inability to abstain from any topical ocular treatments other than unpreserved artificial tears for the duration of the trial
21. Use of autologous serum eye drops (ASED) if started within 2 weeks before the Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
The primary safety endpoint is adverse events' frequency, severity, and duration. | Will be evaluated through study completion (6 weeks)
  Main Adverse Event that will be focused on during the study:
  Irritation and local discomfort Increased Lacrimation Increased mucus Intraocular inflammation Ocular redness Eyelid Edema Hyperemia conjunctival erythema Keratitis
The number of Participants with Treatment-Related Adverse Events | Will be evaluated through study completion (6 weeks)
  as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Patient Tolerability | Will be evaluated through study completion (6 weeks)
  the number of patients discontinuing the study due to plug discomfort.
Plug retention rate | Study termination visit: 6 weeks after plug insertion
  Total patients with plugs remained (did not drop out or lost during the study) at study termination / Total patients with successful plug insertions at Baseline *100
Exploratory Endpoint1 | Will be evaluated from baseline to follow up visit 6 (4 weeks from plug insertion)
  Change from baseline in the study eye in Dryness VAS. The change of measurements from baseline will also be compared between the study and fellow control eye.
Exploratory Endpoint2 | Will be evaluated from baseline to follow up visit 6 (4 weeks from plug insertion)
  Change from baseline in the study eye in CFS. The change of measurements from baseline will also be compared between the study and fellow control eye.
Exploratory Endpoint3 | Will be evaluated from baseline to follow up visit 6 (4 weeks from plug insertion)
  Change from baseline in the study eye in *Schirmer test. The change of measurements from baseline will also be compared between the study and fellow control eye.
  * Change in Schirmer test score would also be compared in visit 3
Exploratory Endpoint4 | Will be evaluated from baseline to follow up visit 6 (4 weeks from plug insertion)
  Change from baseline in the study eye in Lissamine green staining. The change of measurements from baseline will also be compared between the study and fellow control eye.
Exploratory Endpoint5 | Will be evaluated from baseline to termination visit (6 weeks from plug insertion)
  Change from baseline in the study eye in Dryness VAS. The change of measurements from baseline will also be compared between the study and fellow control eye.
Exploratory Endpoint6 | Will be evaluated from baseline to termination visit (6 weeks from plug insertion)
  Change from baseline in the study eye in CFS. The change of measurements from baseline will also be compared between the study and fellow control eye.
Exploratory Endpoint7 | Will be evaluated from baseline to termination visit (6 weeks from plug insertion)
  Change from baseline in the study eye in *Schirmer test score. The change of measurements from baseline will also be compared between the study and fellow control eye.
  * Change in Schirmer test score would also be compared in visit 3
Exploratory Endpoint8 | Will be evaluated from baseline to termination visit (6 weeks from plug insertion)
  Change from baseline in the study eye in Lissamine green staining. The change of measurements from baseline will also be compared between the study and fellow control eye.

CONTACTS AND LOCATIONS:
Overall Officials: Nallely Ramos Betancourt, Dr., Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociación para Evitar la Ceguera en México (APEC), Mexico City, Coyoacán, Mexico

REFERENCES:
- [Background] Baldo A, Cafiero M, Di Caterino P, Di Costanzo L. Tacrolimus ointment in the management of atopic dermatitis. Clin Cosmet Investig Dermatol. 2009 Jan 27;2:1-7. doi: 10.2147/ccid.s3378. PMID 21436963
- [Background] Berdoulay A, English RV, Nadelstein B. Effect of topical 0.02% tacrolimus aqueous suspension on tear production in dogs with keratoconjunctivitis sicca. Vet Ophthalmol. 2005 Jul-Aug;8(4):225-32. doi: 10.1111/j.1463-5224.2005.00390.x. PMID 16008701
- [Background] Ebihara N, Ohashi Y, Fujishima H, Fukushima A, Nakagawa Y, Namba K, Okamoto S, Shoji J, Takamura E, Uchio E, Miyazaki D. Blood level of tacrolimus in patients with severe allergic conjunctivitis treated by 0.1% tacrolimus ophthalmic suspension. Allergol Int. 2012 Jun;61(2):275-82. doi: 10.2332/allergolint.11-OA-0349. Epub 2012 Feb 25. PMID 22361511
- [Result] Fukushima A, Ohashi Y, Ebihara N, Uchio E, Okamoto S, Kumagai N, Shoji J, Takamura E, Nakagawa Y, Namba K, Fujishima H, Miyazaki D. Therapeutic effects of 0.1% tacrolimus eye drops for refractory allergic ocular diseases with proliferative lesion or corneal involvement. Br J Ophthalmol. 2014 Aug;98(8):1023-7. doi: 10.1136/bjophthalmol-2013-304453. Epub 2014 Apr 2. PMID 24695688
- [Result] Haddad EM, McAlister VC, Renouf E, Malthaner R, Kjaer MS, Gluud LL. Cyclosporin versus tacrolimus for liver transplanted patients. Cochrane Database Syst Rev. 2006 Oct 18;2006(4):CD005161. doi: 10.1002/14651858.CD005161.pub2. PMID 17054241
- [Result] Hanifin JM, Paller AS, Eichenfield L, Clark RA, Korman N, Weinstein G, Caro I, Jaracz E, Rico MJ; US Tacrolimus Ointment Study Group. Efficacy and safety of tacrolimus ointment treatment for up to 4 years in patients with atopic dermatitis. J Am Acad Dermatol. 2005 Aug;53(2 Suppl 2):S186-94. doi: 10.1016/j.jaad.2005.04.062. PMID 16021174
- [Result] Kanellopoulos AJ, Asimellis G. In pursuit of objective dry eye screening clinical techniques. Eye Vis (Lond). 2016 Jan 18;3:1. doi: 10.1186/s40662-015-0032-4. eCollection 2016. PMID 26783543
- [Result] Moscovici BK, Holzchuh R, Chiacchio BB, Santo RM, Shimazaki J, Hida RY. Clinical treatment of dry eye using 0.03% tacrolimus eye drops. Cornea. 2012 Aug;31(8):945-9. doi: 10.1097/ICO.0b013e31823f8c9b. PMID 22511024
- [Result] Reitamo S, Ortonne JP, Sand C, Cambazard F, Bieber T, Folster-Holst R, Vena G, Bos JD, Fabbri P, Groenhoej Larsen C; European Tacrolimus Ointment Study Group. A multicentre, randomized, double-blind, controlled study of long-term treatment with 0.1% tacrolimus ointment in adults with moderate to severe atopic dermatitis. Br J Dermatol. 2005 Jun;152(6):1282-9. doi: 10.1111/j.1365-2133.2005.06592.x. PMID 15948994
- See also: Treatment of Dry Eye Using 0.03% Tacrolimus Eye Drops — https://clinicaltrials.gov/ct2/show/NCT01850979
- See also: EagleVision Procedure Demo — https://www.katena.com/education/videos/eaglevision-procedure-demo